CLINICAL TRIAL: NCT04608201
Title: Evaluation of the Efficacy of Nicotine Patches in SARS-CoV2 (COVID-19) Infection in Hospitalized Patients
Acronym: NICOVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200529; 2020-003743-28 (EudraCT Number)
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: SARS-COV2
Keywords: SARS-COV2; COVID19; NICOTINE; transdermal patch
MeSH Terms: conditions — COVID-19 | interventions — Nicotine; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NICOTINE transdermal patch (Experimental): NICOTINE 7 mg / 24h, transdermal patch
  Interventions: Drug: Nicotine 7 mg/ 24h Transdermal Patch - 24 Hour
- Placebo of NICOTINE transdermal patch (Placebo Comparator): Placebo of nicotine patch
  Interventions: Drug: Placebo of NICOTINE Transdermal patch

INTERVENTIONS:
Drug: Nicotine 7 mg/ 24h Transdermal Patch - 24 Hour — Treatment involves escalating doses to the target dose of 14 mg / day
  1. / Dose escalation:
     * Level 1: 3.5 mg/day (1/2 patch) for 2 days (D1 and D2)
     * Level 2: 7 mg/day (1 patch) for 2 days (D3 and D4)
     * Level 3: 10.5 mg/day (1.5 patch) for 2 days (D5 and D6)
     * Level 4: target dose = 14 mg/day (from D7 to discharge from hospital + 1 week or maximum 5 weeks after the start of treatment)
  2. / Decrease in dose (1 week after exit from hospital or maximum 5 weeks after the start of treatment): Decrease of 3.5 mg (1/2 patch) per week (over 3 weeks maximum)
  Arms: NICOTINE transdermal patch
Drug: Placebo of NICOTINE Transdermal patch — Placebo of nicotine patch administered to the same administration schedule as in the experimental arm
  Arms: Placebo of NICOTINE transdermal patch

SUMMARY:
The coronavirus disease (COVID-19) epidemic represents a major therapeutic challenge. The highly contagious severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) and the long duration of the disease have led to a massive influx of patients admitted in health services and intensive care units. To current knowledge, there is no treatment yet that that can prevent infection from SARS-COV-2 virus, nor the disease progression to a severe form.

Daily active smokers are rare among outpatients or hospitalized COVID-19 patients.

Several arguments suggest that nicotine could be responsible for this protective effect thank to the nicotinic acetylcholine receptor (nAChR).

Based on epidemiological data and experimental data from scientific literature, we hypothesize that nicotine could inhibit the penetration and spread of the virus and improve the management of COVID19 , particularly in hospitalized patients to prevent adverse outcomes (death, transfer to intensive care unit, care limitation, mechanical ventilation an high flow oxygen).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients hospitalized for less than 72 hours
* Non-smoking and non-vaping patients (for former smokers or former vapers: abstinent for at least 12 months)
* Documented diagnosis of COVID19
* Lung disease suggestive of COVID-19 on chest scanner or need for oxygen therapy
* Obtaining, informed and signed consent
* Affiliated to a social security scheme or beneficiary of such a scheme (except AME)

Exclusion Criteria:

* WHO 10-point Clinical Progression Scale score > 5 (patient on non-invasive or mechanical ventilation, patient in need of high-flow oxygen therapy)
* Indication of transfer to intensive care unit (oxygen therapy> 8 L / min ; out or not carried out due to LATA)
* Current treatment with nicotine replacement therapy, bupropion or varenicline in the last 30 days
* Known addiction problem to alcohol or other substances
* Contraindication for nicotine patches:

  * pregnant or breastfeeding woman
  * lack of effective contraception for women of childbearing age
  * Generalized skin pathologies that may interfere with the use of a transdermal patch
  * stroke or myocardial infarction or acute coronary syndrome for less than 3 months
  * allergy to nicotine or to one of the excipients of the transdermal patch
  * Uncontrolled high blood pressure
  * Unstable or worsening angina
  * Severe cardiac arrhythmia (defined by wearing an automatic implantable defibrillator)
  * Known obliterating peripheral arterial disease
  * Known severe heart failure with an ejection fraction <30%)
  * Known severe renal (ClCr <30 ml / min) or hepatic (Child C) impairment
  * Known pheochromocytoma
  * Known uncontrolled hyperthyroidism
  * Esophagitis due to gastroesophageal reflux disease or an active peptic ulcer
* Patient included in another interventional trial evaluating a health product
* Patient under guardianship or curatorship
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
The unfavorable outcome on Day 14 | Day 14
  Defined by scores higher than 5 on the World Health Organization 10-point Clinical Progression Scale (WHO-CPS) on day 14

SECONDARY OUTCOMES:
Survival rate | Day 14, Day 28
Proportion of transfer to intensive care unit (ICU) | Day 14, Day 28
Proportion of indication of transfer to intensive care unit (carried out or not in case of LATA) | Day 14, Day 28
Number of days living without mechanical ventilation | Day 14, Day 28
Number of days living without non-invasive ventilation and mechanical ventilation | Day 4, Day 14, Day 28
Proportion of patient with a score higher than 6 on the World Health Organization 10-point Clinical Progression Scale | Day 14
Duration of hospitalization | Fom day 1 up to 3 month
Proportion of patient in each category of the World Health Organization 10-point Clinical Progression Scale | Day 7, Day 14 and Day 28
Proportion of patient in each category of the National Early Warning Scale (NEWS) 2 | Day 7, Day14 and Day28 (or the day of discharge from hospital)
Proportion of patient with a SARS-CoV-2 viral load detection | Day 7 or the day of discharge from hospital if before day 7
Mean evolution of blood count | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of platelets | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of blood ionogram | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of glycemia | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of serum creatinine | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of C reactive protein | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of Interleukin 6 (IL-6) | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of oxygen requirements (number of liters / min) | At randomization then every 3 days until discharge, or up to 5 weeks
Mean evolution of SaO2 | At randomization then every 3 days until discharge, or up to 5 weeks
Proportion of active smoker or active vapers or taking nicotine substitutes documented by examination | Week 2 after treatment decrease, Week 8 after treatment decrease
Proportion of active smoker or active vapers or taking nicotine substitutes documented by urinary cotinine | Week 8 after treatment decrease
Mean score of Desire to smoke defined by French Tobacco Craving questionnaire (FTCQ12 ) | Week 2 after treatment decrease, Week 8 after treatment decrease
Mean score of Cigarette Withdrawal Scale (CWS) | Week 2 after treatment decrease, Week 8 after treatment decrease
Mean score of Hospital anxiety and depression scale (HAD) | Week 2 after treatment decrease, Week 8 after treatment decrease
Mean score of Positive and Negative Affect Schedule (PANAS) | Week 2 after treatment decrease, Week 8 after treatment decrease
Mean score of Insomnia severity scale (ISI) | Week 2 after treatment decrease, Week 8 after treatment decrease
weight evolution | Day 1, Week 2 after treatment decrease, Week 8 after treatment decrease

CONTACTS AND LOCATIONS:
Overall Officials: Valérie POURCHER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Pitié-Salpêtrière - AP-HP, Paris, France